CLINICAL TRIAL: NCT05129397
Title: A Randomized Controlled Trial to Improve Biobehavioral Regulation Among High-Adversity Mothers and Young Children
Brief Title: Virtual Mom Power With High-Adversity Mothers and Children (MPHAMC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sarah Gray, Associate Professor of Psychology, Clinical Professor of Psychiatry & Behavioral Sciences, Principal Investigator, Tulane University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-2012-TU Uptown; K23MH119047 (NIH)
Record Dates: First submitted 2021-10-25; First posted 2021-11-22 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Psychopathology
Keywords: biobehavioral regulation; Respiratory Sinus Arrhythmia; parenting behavior
MeSH Terms: conditions — Arrhythmia, Sinus

STUDY DESIGN:
Intervention Model Description: There are two arms: an experimental group receiving the Mom Power group intervention over 10 weeks, and a control group that will receive informational virtual mailings over 10 weeks. Treatment delivery will be consistent with the Mom Power manual and informational mailings will contain content from the Mom Power Curriculum.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The experimental arm of Virtual Mom Power is a manualized multi-family group intervention consisting of 10, 90-minute virtual group + 2 individual sessions led by two co-facilitators. The curriculum includes 5 core components: (1) Attachment-Focused Parenting Education; (2) Self-Care; (3) Parenting Practice; (4) Social Support; & (5) Connection to Resources. Individual sessions combine motivational interviewing with MP core components and focus on identifying goals and barriers. We will work with mothers in individual coaching to problem-solve childcare and privacy during group time. Weekly between-group phone/text check-ins are also a part of the curriculum, used to strengthen connection, build trust, ensure safety, and assess basic needs. Data regarding attendance will be recorded and total dosage examined in treatment effects.
  Interventions: Behavioral: Mom Power
- Informational control (Active Comparator): The control arm of this study consists of two individual sessions with mothers, along with 10 weeks of virtual informational mailings. The mailings will contain Mom Power curriculum about attachment-based parenting and self-care. The individual sessions will focus on individual goal-setting related to parenting and reflection on the parent-child relationship. The control group does not include the components of social support, affect regulation skills coaching, or guided parent-child interaction that are part of the experimental arm.
  Interventions: Behavioral: Mom Power Informational Mailing

INTERVENTIONS:
Behavioral: Mom Power — Virtual Mom Power is a manualized multi-family group intervention consisting of 10 virtual group + 2 individual sessions led by two masters-level co-facilitators. Virtual groups are 90 minutes, following a structured format via secure HIPAA compatible video platform. The curriculum includes 5 core components: (1) Attachment-Focused Parenting Education; (2) Self-Care; (3) Parenting Practice (4) Social Support; & (5) Connection to Resources. Individual sessions combine motivational interviewing with MP core components and focus on identifying goals and barriers. Weekly between-group phone/text check-ins are also a part of the curriculum, used to strengthen connection, build trust, ensure safety, and assess basic needs.
  Arms: Treatment
Behavioral: Mom Power Informational Mailing — This active comparison condition intervention includes two individual sessions along with 10 weeks of informational mailing with content related to Mom Power core concepts.
  Arms: Informational control

SUMMARY:
This study is a randomized controlled confirmatory efficacy trial of virtual Mom Power (MP), a group-based, relationship-focused multifamily preventive intervention.

DETAILED DESCRIPTION:
This study is a randomized controlled confirmatory efficacy trial of virtual Mom Power (MP), a group-based, relationship-focused multifamily intervention with previously demonstrated effectiveness improving maternal mental health and parenting stress in randomized controlled trials. vMP targets 5 core components: 1) enhancing social support; 2) attachment-based parenting education; 3) self-care, including affect regulation; 4) guided parent-child interactions, and 5) connecting to care. Eligible and enrolled participants will be randomized to receive the 10 week group-based intervention or 10 weeks of informational mailings; both groups will receive individual home-based sessions. Outcomes include maternal social support, psychopathology, sensitive parenting, child psychopathology, two-generational biobehavioral self-regulation targets (Respiratory Sinus Arrhythmia), parent and child emotion and behavior regulation, and dyadic behavioral and physiological synchrony. Assessments will occur at intake, post, and 6 months following the group.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment status in one of the following services: Supplemental Nutrition Assistance Program (SNAP), Family Independence Temporary Assistance Program (FITAP), Medicaid, Special Supplemental Nutrition Program for Women, Infants, and Children (WIC), or Head Start
* Maternal age of at least 18 years
* Mother is primary caregiver of child
* Mother speaks English
* Child age is between 3-5 years
* Family resides within 8 parish New Orleans metro area

Exclusion Criteria:

* Mother is not biological mother
* Diagnosis of a heart condition in the mother or the child
* Presence of a pacemaker in the mother or the child
* Child diagnosis of autism or global developmental delay
* Active maternal substance use
* Active maternal psychosis

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only biological mothers are eligible to participate due to concerns about heritability of physiological outcomes. Children of all sexes are eligible.
Enrollment: 44 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline maternal depressive symptoms at post-intervention | At completion of intervention, approximately 3 months
  Mothers will report on their own depressive symptoms using the Patient Health Questionnaire-9 (PHQ-9) at baseline, post-intervention, and 6 month follow up; change in sum scale from baseline at post-intervention will be assessed. Higher scores reflect more depressive symptoms.
Change from baseline maternal depressive symptoms at 6 month follow up | 6 months (follow up)
  Mothers will report on their own depressive symptoms using the Patient Health Questionnaire-9 (PHQ-9) at baseline, post-intervention, and 6 month follow up; change in sum scale from baseline to 6 month follow up will be assessed. Higher scores reflect more depressive symptoms.
Change from baseline maternal posttraumatic stress symptoms at post-intervention | At completion of intervention, approximately 3 months
  Mothers will report on their own posttraumatic stress symptoms using the Posttraumatic Checklist for Diagnostic and Statistical Manual Diploma in Social Medicine-5 (PCL-5). Sum scales will be assessed at baseline, post-intervention (3 months), and 6 month follow up; change in sum scale from baseline to 3 month follow up will be assessed. Higher scores reflect more posttraumatic stress symptoms.
Change from baseline maternal posttraumatic stress symptoms at 6 month follow up | 6 months (follow up)
  Mothers will report on their own posttraumatic stress symptoms using the Posttraumatic Checklist for Diagnostic and Statistical Manual Diploma in Social Medicine-5 (PCL-5). Sum scales will be assessed at baseline, post-intervention (3 months), and 6 month follow up; change in sum scale from baseline to 6 month follow up will be assessed. Higher scores reflect more posttraumatic stress symptoms.
Change from baseline child behavior at post-intervention | At completion of intervention, approximately 3 months
  Mothers will report on child behavior on the Child Behavior Checklist (CBCL 1.5-5). Sum scores will be used. Higher scores reflect more behavior problems.
Change from baseline child behavior at 6 month follow up. | 6 months (follow up)
  Mothers will report on child behavior on the Child Behavior Checklist (CBCL 1.5-5). Sum scores will be used. Higher scores reflect more behavior problems.

SECONDARY OUTCOMES:
Change in parenting stress from baseline to post-intervention | At completion of intervention, approximately 3 months
  Mothers will report on their own parenting stress using the Parenting Stress Index - 4, Short Form (PSI-SF); change in the the Total Stress scale from baseline to post-assessment (3 months) will be examined. Higher scores reflect more parenting stress.
Change in parenting stress from baseline to 6 month follow up | 6 months
  Mothers will report on their own parenting stress using the Parenting Stress Index - 4, Short Form (PSI-SF); change in the the Total Stress scale from baseline to follow up (6 months) will be examined. Higher scores reflect more parenting stress.
Change in self-report parent child relationship from baseline to post intervention | At completion of intervention, approximately 3 months
  Mothers will report on their own parenting stress using the Parenting Stress Index - 4, Short Form (PSI-SF); change in the the Parent Child Dysfunctional Interaction scale from baseline to post-assessment (3 months) will be examined. Higher scores reflect more dysfunction.
Change in self-report parent child relationship from baseline to follow up | 6 months
  Mothers will report on their own parenting stress using the Parenting Stress Index - 4, Short Form (PSI-SF); change in the the Parent Child Dysfunctional Interaction scale from baseline to follow up (6 months) will be examined. Higher scores reflect more dysfunction.
Change in maternal social support from baseline to post intervention | At completion of intervention, approximately 3 months
  Mothers will report on their perceived social support a using the Multidimensional Scale of Perceived Social Support (MSPSS). Change from baseline to post intervention (3 months) will be examined. Higher scores reflect more social support.
Change in maternal social support from baseline to follow up | 6 months
  Mothers will report on their perceived social support a using the Multidimensional Scale of Perceived Social Support (MSPSS). Change from baseline to follow up (6 months) will be examined. Higher scores reflect more social support.
Change in observed parenting sensitivity from baseline to post-intervention | At completion of intervention, approximately 3 months
  Parenting sensitivity will be assessed at baseline and post intervention (3 months) with an observational measure. Video tapes of parent-child interactions during a 5-minute period of free play and a 5-minute period of structured interaction with a challenging puzzle will be coded using the Coding Interactive Behavior (CIB) measure. Parenting sensitivity scales will be used. Higher scores reflect more sensitivity.
Change in Working Models from baseline to post-intervention | At completion of intervention, approximately 3 months
  Mothers and evaluators will complete a Working Model of the Child Interview (WMCI) at baseline and post-intervention (3 months) to assess parents' internal working model classifications. Classifications as Balanced, Disengaged, and Distorted will be used. Classification as balance is considered a more adaptive outcome.
Change in maternal emotion regulation from baseline to post-intervention | At completion of intervention, approximately 3 months
  Mothers will report on their difficulties in emotion regulation (Difficulties in Emotion Regulation Scale). Change in the sum score from baseline to post-intervention will be examined. Higher scores reflect more difficulties in emotion regulation.
Change in maternal emotion regulation from baseline to follow up | 6 months
  Mothers will report on their difficulties in emotion regulation (Difficulties in Emotion Regulation Scale). Change in the sum score from baseline to 6 month follow up will be examined. Higher scores reflect more difficulties in emotion regulation.
Change in maternal emotion regulation while parenting from baseline to post intervention | At completion of intervention, approximately 3 months
  Mothers will report on their parenting-specific behavioral self-regulation (Regulating Emotions in Parenthood). Change in the sum score from baseline to post intervention will be examined.
Change in maternal emotion regulation while parenting from baseline to follow up | 6 months
  Mothers will report on their parenting-specific behavioral self-regulation (Regulating Emotions in Parenthood). Change in the sum score from baseline to 6 month follow up will be examined.
Change in maternal resting Respiratory Sinus Arrhythmia from baseline to post-intervention | At completion of intervention, approximately 3 months
  At baseline assessments and at post-intervention assessments, electrocardiogram data will be collected during a 2 minute neutral video tsak. ECG signals will be synchronized at acquisition with video and processed offline using Mindware software; research assistants will visually inspect for missing or erroneously identified R-peaks. Using spectral analysis of interbeat intervals, high-frequency heart rate variability will be extracted to quantify respiratory sinus arrhythmia (RSA) within frequency bandwidths associated with respiration (.15-.40 for mothers) and log-transformed. Change in resting RSA from baseline to post-intervention will be examined. Higher resting RSA is expected post-intervention.
Change in maternal Respiratory Sinus Arrhythmia reactivity from baseline to post-intervention | At completion of intervention, approximately 3 months
  Electrocardiogram data will be collected during a 2 minute baseline neutral video task and a 5 minute parent-child puzzle teaching task. ECG signals will be synchronized at acquisition with video and processed offline using Mindware software; research assistants will visually inspect for missing or erroneously identified R-peaks. Using spectral analysis of interbeat intervals, high-frequency heart rate variability will be extracted to quantify RSA within frequency bandwidths associated with respiration (24-1.04 for children) and log-transformed. Respiratory Sinus Arrhythmia reactivity in response to the puzzle task will be assessed at baseline and post-intervention (3 months)
Change in child resting Respiratory Sinus Arrhythmia from baseline to post-intervention | At completion of intervention, approximately 3 months
  Electrocardiogram data will be collected during a 2 minute baseline neutral video task. ECG signals will be synchronized at acquisition with video and processed offline using Mindware software; research assistants will visually inspect for missing or erroneously identified R-peaks. Using spectral analysis of interbeat intervals, high-frequency heart rate variability will be extracted to quantify RSA within frequency bandwidths associated with respiration (24-1.04 for children) and log-transformed. Change in children's resting Respiratory Sinus Arrhythmia during the neutral task will be assessed from baseline to post-intervention (3 months). Higher resting RSA is expected post-intervention.
Change in child Respiratory Sinus Arrhythmia reactivity from baseline to post-intervention | At completion of intervention, approximately 3 months
  Electrocardiogram data will be collected during a 2 minute baseline neutral video task and a 5 minute parent-child puzzle teaching task. ECG signals will be synchronized at acquisition with video and processed offline using Mindware software; research assistants will visually inspect for missing or erroneously identified R-peaks. Using spectral analysis of interbeat intervals, high-frequency heart rate variability will be extracted to quantify RSA within frequency bandwidths associated with respiration (24-1.04 for children) and log-transformed. Change in children's Respiratory Sinus Arrhythmia reactivity during the puzzle task from baseline to post-intervention will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Gray, PhD, Principal Investigator — Tulane University
Locations (1):
- Tulane Child and Family Lab, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lowe B, Unutzer J, Callahan CM, Perkins AJ, Kroenke K. Monitoring depression treatment outcomes with the patient health questionnaire-9. Med Care. 2004 Dec;42(12):1194-201. doi: 10.1097/00005650-200412000-00006. PMID 15550799
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Achenbach, T. M., & Rescorla, L. A. (2000). Manual for the ASEBA preschool forms & profiles: An integrated system of multi-informant assessment. University of Vermont.
- [Background] Abidin, Richard R. Parenting stress index-short form. Charlottesville, VA: Pediatric psychology press, 1990.
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Feldman R, Granat A, Pariente C, Kanety H, Kuint J, Gilboa-Schechtman E. Maternal depression and anxiety across the postpartum year and infant social engagement, fear regulation, and stress reactivity. J Am Acad Child Adolesc Psychiatry. 2009 Sep;48(9):919-927. doi: 10.1097/CHI.0b013e3181b21651. PMID 19625979
- [Background] Zeanah, C. H. (2007). Constructing a relationship formulation for mother and child: Clinical application of the Working Model of the Child Interview. In D. Oppenheim & D. F. Goldsmith (Eds.), Attachment Theory in Clinical Work with Children: Bridging the Gap Between Research and Practice (pp. 3-30). New York, NY: Guilford Press.
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment, 26(1), 41-54
- [Background] Rodriguez VJ, Shaffer A. Validation of the Regulating Emotions in Parenting Scale (REPS): Factor structure and measurement invariance. J Fam Psychol. 2021 Jun;35(4):468-477. doi: 10.1037/fam0000808. Epub 2020 Sep 17. PMID 32940490
- [Background] Conduct Problems Prevention Research Group. Initial impact of the Fast Track prevention trial for conduct problems: I. The high-risk sample. Conduct Problems Prevention Research Group. J Consult Clin Psychol. 1999 Oct;67(5):631-47. PMID 10535230
- [Background] Smith-Donald, R., Raver, C. C., Hayes, T., & Richardson, B. (2007). Preliminary construct and concurrent validity of the Preschool Self-regulation Assessment (PSRA) for field-based research. Early Childhood Research Quarterly, 22(2), 173-187
- [Background] Rosenblum KL, Muzik M, Morelen DM, Alfafara EA, Miller NM, Waddell RM, Schuster MM, Ribaudo J. A community-based randomized controlled trial of Mom Power parenting intervention for mothers with interpersonal trauma histories and their young children. Arch Womens Ment Health. 2017 Oct;20(5):673-686. doi: 10.1007/s00737-017-0734-9. Epub 2017 Jun 25. PMID 28647759
- [Background] Rosenblum K, Lawler J, Alfafara E, Miller N, Schuster M, Muzik M. Improving Maternal Representations in High-Risk Mothers: A Randomized, Controlled Trial of the Mom Power Parenting Intervention. Child Psychiatry Hum Dev. 2018 Jun;49(3):372-384. doi: 10.1007/s10578-017-0757-5. PMID 28936602